CLINICAL TRIAL: NCT07147764
Title: Comparison of the Effect of Pain Neuroscience Education Combined With Physiotherapy, and Physiotherapy Alone in Temporomandibular Disorders
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ainaz Shahedi (Other)
Collaborators: Medipol University (Other)
Responsible Party: Sponsor-Investigator, Ainaz Shahedi, MSc Candidate in Physiotherapy, Istanbul Medipol University, Istanbul Medipol University Hospital
Organization: Istanbul Medipol University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E-10840098-202.3.02-2936
Record Dates: First submitted 2025-08-22; First posted 2025-08-29 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Temporomandibular Joint Disorders
Keywords: Temporomandibular Disorder; Pain Neuroscience Education; Chronic Pain
MeSH Terms: conditions — Temporomandibular Joint Disorders; Chronic Pain | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (CG): Physiotherapy (Active Comparator)
  Interventions: Other: Physiotherapy
- Pain Neuroscience Group (PNEG): Physiotherapy + Pain Neuroscience Education (Experimental)
  Interventions: Behavioral: Pain Neuroscience Education

INTERVENTIONS:
Other: Physiotherapy — Physiotherapy treatment programs include therapeutic ultrasound, muscle relaxation techniques, range of motion exercises, and joint and soft tissue mobilization.
  Arms: Control group (CG): Physiotherapy
Behavioral: Pain Neuroscience Education — PNE sessions will be conducted in addition to physiotherapy programs for intervention groups. PNE sessions will occupy half of each session during the first two weeks. Physiotherapists trained in PNE will deliver sessions using a combination of metaphors, animated videos, and scientifically accurate descriptions. The same physiotherapist will lead both sessions with the same patient.
  Active learning techniques will include:
  Connecting new information with prior knowledge. Operationalizing key pain concepts into individual contexts. Facilitated problem-solving and critical reflection.
  Arms: Pain Neuroscience Group (PNEG): Physiotherapy + Pain Neuroscience Education

SUMMARY:
This research study aims to evaluate the effectiveness of Pain Neuroscience Education (PNE) when it is added to a physiotherapy program for people experiencing chronic temporomandibular disorders (TMD). To see whether adding PNE to physiotherapy program would provides additional benefits in reducing pain intensity, improving psychological well-being, and enhancing functional outcomes. The findings are expected to provide new insights into more comprehensive and patient-centered treatment strategies for managing chronic TMD.

Participants will be randomly assigned to one of two groups:

Control Group: Physiotherapy only

PNE Group: Physiotherapy plus Pain Neuroscience Education

Both groups will receive their respective treatments for a set period of time.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with pain-related TMDs according to DC/TMD guidelines
* Chronic TMD pain, defined as experiencing pain for at least six months and feeling the pain during the last 30 days
* Age between 18-65 years

Exclusion Criteria:

* Illiterate patients
* Severe depression (medical diagnoses)
* Previous diagnosis of uncontrolled psychiatric disorder neurodegenerative diseases
* Clinical history of tumors in the craniofacial region
* Patients in the post dental surgery period
* Patients who were submitted to previous physical therapy in the past year or to any health/pain education strategy
* Pregnant women
* Infections, whiplash-associated disorders and with chronic degenerative inflammatory or neurologic disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-09-14 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
The Craniofacial Pain and Disability Inventory (CF-PDI) | Baseline, 1 month after start of treatment, Immediate post-treatment, 3 month follow up
  It consists of 21 items, with a score ranging from 0 to 63 points. Each question is scored on a 4-point ordinal scale, ranging from 0 to 3. A higher score reflects higher disability levels.

SECONDARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | Baseline, 1 month after start of treatment, Immediate post-treatment, 3 month follow up
  It includes an 11-point numerical rating scale, ranging from 0, indicating (no pain), to 10, representing (the worst pain imaginable),.
Pain Self-Efficacy Questionnaire (PSEQ) | Baseline, 1 month after start of treatment, Immediate post-treatment, 3 month follow up
  It consists of 10 items scored on a 7-point ordinal scale (ranging from 0: "not at all confident" to 6: "completely confident").
Pain Catastrophizing Scale (PCS) | Baseline,1 month after start of treatment, Immediate post-treatment, 3 month follow up
  It consists of 13 items for the assessment of catastrophizing thoughts. It is divided into three domains: helplessness, magnification, and rumination. Each item is scored on a 5-point ordinal scale. The PCS total score ranges from 0 to 52 points, higher values denote greater pain catastrophizing.
Hospital Anxiety and Depression Scale (HADS) | Baseline, 1 month after start of treatment, Immediate post-treatment, 3 month follow up
  It comprises two subscales: HADS-Anxiety (HADS-A) and HADS-Depression (HADS-D), each consisting of seven items distributed throughout the questionnaire. Every item is rated on a 4-point Likert scale ranging from 0 to 3, reflecting the severity of symptoms. A score of 8 or above on either subscale is considered indicative of possible anxiety or depression.
The Tampa Scale for Kinesiophobia specific to Temporomandibular Disorders (TSK-TMD) | Baseline, 1 month after start of treatment, Immediate post-treatment, 3 month follow up
  It consists of 12 items. Each item is scored on a 4-point ordinal scale, ranging from "strongly disagree" (score = 1) to "strongly agree" (score = 4). Ratings are summed to yield a total score. Higher scores reflect a greater fear of movement (12-48 points).
Revised Neurophysiology of Pain Questionnaire (rNPQ) | Baseline, 1 month after start of treatment, Immediate post-treatment, 3 month follow up
  It includes 12 items, each requiring a true, false, or undecided response. Each correct answer receives one point, while incorrect or undecided answers receive zero. Total scores range from 0 to 12, with higher scores reflecting greater knowledge of pain-related physiological concepts.
The Exercise Adherence Rating Scale (EARS) | Baseline, 1 month after start of treatment, Immediate post-treatment, 3 month follow up
  The tool consists of six items rated on a five-point Likert scale, ranging from 0 (strongly agree) to 4 (totally disagree). Items with positively worded statements are reverse-scored to maintain consistency in interpretation. The total adherence score ranges from 0 to 24, with higher scores indicating greater adherence to the exercise regimen.
Fear Avoidance Components Scale (FACS) | Baseline, 1 month after start of treatment, Immediate post-treatment, 3 month follow up
  This self-administered questionnaire comprises 20 items rated on a 6-point Likert scale, ranging from 0 (completely disagree) to 6 (completely agree), yielding a maximum score of 100. Higher scores indicate stronger fear-avoidance beliefs.

CONTACTS AND LOCATIONS:
Overall Officials: Gizem Ergezen Şahin, Dr. Assistant Professor, Study Director — Department of Physiotherapy and Rehabilitation/Istanbul Medipol University
Locations (1):
- Istanbul Medipol University, Istanbul, Kavacik, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
At present, there is no plan to share individual participant data (IPD) outside the research team due to the small sample size and confidentiality considerations. However, in the future, de-identified data may be shared if required by institutional policy, journal requirements, or upon reasonable request from qualified researchers, always in accordance with ethical and legal standards.

REFERENCES:
- [Background] Justribo-Manion C, Mesa-Jimenez J, Bara-Casaus J, Zuil-Escobar JC, Wachowska K, Alvarez-Bustins G. Additional effects of therapeutic exercise and education on manual therapy for chronic temporomandibular disorders treatment: a randomized clinical trial. Physiother Theory Pract. 2025 Jan;41(1):12-27. doi: 10.1080/09593985.2024.2316305. Epub 2024 Feb 14. PMID 38353484
- [Background] von Piekartz H, Bleiss S, Herzer S, Hall T, Ballenberger N. Does combining oro-facial manual therapy with bruxism neuroscience education affect pain and function in cases of awake bruxism? A pilot study. J Oral Rehabil. 2024 Sep;51(9):1692-1700. doi: 10.1111/joor.13740. Epub 2024 Jun 18. PMID 38894567
- [Background] Wood L, Hendrick PA. A systematic review and meta-analysis of pain neuroscience education for chronic low back pain: Short-and long-term outcomes of pain and disability. Eur J Pain. 2019 Feb;23(2):234-249. doi: 10.1002/ejp.1314. Epub 2018 Oct 14. PMID 30178503
- [Background] Kasimis K, Apostolou T, Kallistratos I, Lytras D, Iakovidis P. Effects of Manual Therapy Plus Pain Neuroscience Education with Integrated Motivational Interviewing in Individuals with Chronic Non-Specific Low Back Pain: A Randomized Clinical Trial Study. Medicina (Kaunas). 2024 Mar 29;60(4):556. doi: 10.3390/medicina60040556. PMID 38674202
- [Background] Babatunde OO, Jordan JL, Van der Windt DA, Hill JC, Foster NE, Protheroe J. Effective treatment options for musculoskeletal pain in primary care: A systematic overview of current evidence. PLoS One. 2017 Jun 22;12(6):e0178621. doi: 10.1371/journal.pone.0178621. eCollection 2017. PMID 28640822
- [Background] Lin I, Wiles L, Waller R, Goucke R, Nagree Y, Gibberd M, Straker L, Maher CG, O'Sullivan PPB. What does best practice care for musculoskeletal pain look like? Eleven consistent recommendations from high-quality clinical practice guidelines: systematic review. Br J Sports Med. 2020 Jan;54(2):79-86. doi: 10.1136/bjsports-2018-099878. Epub 2019 Mar 2. PMID 30826805
- [Background] Watson JA, Ryan CG, Cooper L, Ellington D, Whittle R, Lavender M, Dixon J, Atkinson G, Cooper K, Martin DJ. Pain Neuroscience Education for Adults With Chronic Musculoskeletal Pain: A Mixed-Methods Systematic Review and Meta-Analysis. J Pain. 2019 Oct;20(10):1140.e1-1140.e22. doi: 10.1016/j.jpain.2019.02.011. Epub 2019 Mar 1. PMID 30831273
- [Background] Lepri B, Romani D, Storari L, Barbari V. Effectiveness of Pain Neuroscience Education in Patients with Chronic Musculoskeletal Pain and Central Sensitization: A Systematic Review. Int J Environ Res Public Health. 2023 Feb 24;20(5):4098. doi: 10.3390/ijerph20054098. PMID 36901108
- [Background] Louw A, Schuemann T, Zimney K, Puentedura EJ. Pain Neuroscience Education for Acute Pain. Int J Sports Phys Ther. 2024 Jun 2;19(6):758-767. doi: 10.26603/001c.118179. eCollection 2024. PMID 38835986
- [Background] Wadhokar OC, Patil DS. Current Trends in the Management of Temporomandibular Joint Dysfunction: A Review. Cureus. 2022 Sep 19;14(9):e29314. doi: 10.7759/cureus.29314. eCollection 2022 Sep. PMID 36277551
- [Background] Yao L, Sadeghirad B, Li M, Li J, Wang Q, Crandon HN, Martin G, Morgan R, Florez ID, Hunskaar BS, Wells J, Moradi S, Zhu Y, Ahmed MM, Gao Y, Cao L, Yang K, Tian J, Li J, Zhong L, Couban RJ, Guyatt GH, Agoritsas T, Busse JW. Management of chronic pain secondary to temporomandibular disorders: a systematic review and network meta-analysis of randomised trials. BMJ. 2023 Dec 15;383:e076226. doi: 10.1136/bmj-2023-076226. PMID 38101924
- [Background] Urbanski P, Trybulec B, Pihut M. The Application of Manual Techniques in Masticatory Muscles Relaxation as Adjunctive Therapy in the Treatment of Temporomandibular Joint Disorders. Int J Environ Res Public Health. 2021 Dec 8;18(24):12970. doi: 10.3390/ijerph182412970. PMID 34948580
- [Background] Ferrillo M, Giudice A, Marotta N, Fortunato F, Di Venere D, Ammendolia A, Fiore P, de Sire A. Pain Management and Rehabilitation for Central Sensitization in Temporomandibular Disorders: A Comprehensive Review. Int J Mol Sci. 2022 Oct 12;23(20):12164. doi: 10.3390/ijms232012164. PMID 36293017
- [Background] Garstka AA, Kozowska L, Kijak K, Brzozka M, Gronwald H, Skomro P, Lietz-Kijak D. Accurate Diagnosis and Treatment of Painful Temporomandibular Disorders: A Literature Review Supplemented by Own Clinical Experience. Pain Res Manag. 2023 Jan 31;2023:1002235. doi: 10.1155/2023/1002235. eCollection 2023. PMID 36760766
- [Background] Cho YK, Jung YL, Im A, Hong SJ, Kim K. Social Media-Based Pain Neuroscience Education for Temporomandibular Joint Disorder: A Randomized Controlled Trial. Pain Manag Nurs. 2025 Jun;26(3):e261-e269. doi: 10.1016/j.pmn.2024.12.010. Epub 2025 Jan 17. PMID 39827051
- [Background] Li DTS, Leung YY. Temporomandibular Disorders: Current Concepts and Controversies in Diagnosis and Management. Diagnostics (Basel). 2021 Mar 6;11(3):459. doi: 10.3390/diagnostics11030459. PMID 33800948
- [Background] Dos Santos Aguiar A, Bataglion C, Felicio LR, Azevedo B, Chaves TC. Additional effect of pain neuroscience education to craniocervical manual therapy and exercises for pain intensity and disability in temporomandibular disorders: a study protocol for a randomized controlled trial. Trials. 2021 Sep 6;22(1):596. doi: 10.1186/s13063-021-05532-x. PMID 34488856
- [Background] Ferneini EM. Temporomandibular Joint Disorders (TMD). J Oral Maxillofac Surg. 2021 Oct;79(10):2171-2172. doi: 10.1016/j.joms.2021.07.008. No abstract available. PMID 34620421
- [Background] Chimenti RL, Frey-Law LA, Sluka KA. A Mechanism-Based Approach to Physical Therapist Management of Pain. Phys Ther. 2018 May 1;98(5):302-314. doi: 10.1093/ptj/pzy030. PMID 29669091
- [Background] Busse JW, Casassus R, Carrasco-Labra A, Durham J, Mock D, Zakrzewska JM, Palmer C, Samer CF, Coen M, Guevremont B, Hoppe T, Guyatt GH, Crandon HN, Yao L, Sadeghirad B, Vandvik PO, Siemieniuk RAC, Lytvyn L, Hunskaar BS, Agoritsas T. Management of chronic pain associated with temporomandibular disorders: a clinical practice guideline. BMJ. 2023 Dec 15;383:e076227. doi: 10.1136/bmj-2023-076227. PMID 38101929
- [Background] List T, Jensen RH. Temporomandibular disorders: Old ideas and new concepts. Cephalalgia. 2017 Jun;37(7):692-704. doi: 10.1177/0333102416686302. Epub 2017 Jan 9. PMID 28068790
- [Background] Liou YJ, Bai YM, Tsai SJ, Chen TJ, Chen MH, Lo WL. Bidirectional Associations of Temporomandibular Joint Disorders with Major Depressive and Anxiety Disorders. J Evid Based Dent Pract. 2023 Jun;23(2):101860. doi: 10.1016/j.jebdp.2023.101860. Epub 2023 Mar 17. PMID 37201980
- [Background] Al-Jewair T, Shibeika D, Ohrbach R. Temporomandibular Disorders and Their Association with Sleep Disorders in Adults: A Systematic Review. J Oral Facial Pain Headache. 2021 Winter;35(1):41-53. doi: 10.11607/ofph.2780. PMID 33730126
- [Background] A. Aggarwal, J. Gadekar, and P. Kakodkar, "Role of Myofascial Release Technique on Mobility and Function in Temporomandibular Joint Disorder Patients with Neck Pain," J. Dent. Res. Rev., vol. 7, no. Suppl 1, 2020
- [Background] Zielinski G, Pajak-Zielinska B, Ginszt M. A Meta-Analysis of the Global Prevalence of Temporomandibular Disorders. J Clin Med. 2024 Feb 28;13(5):1365. doi: 10.3390/jcm13051365. PMID 38592227
- [Background] McNeill C. Management of temporomandibular disorders: concepts and controversies. J Prosthet Dent. 1997 May;77(5):510-22. doi: 10.1016/s0022-3913(97)70145-8. PMID 9151272